CLINICAL TRIAL: NCT04576182
Title: Investigating Mechanisms of Change in Supportive-Expressive vs. Emotion-Focused Treatment of Depression Using a Personalized Treatment Approach: The Case of the Theories of Weakness vs. Strength
Brief Title: Supportive-Expressive and Emotion-Focused Treatment for Depression
Acronym: SETEFT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Haifa (Other)
Collaborators: Israel Science Foundation (Other)
Responsible Party: Principal Investigator, Sigal Zilcha Mano, Associate Professor, University of Haifa
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ISF 395/19
Record Dates: First submitted 2020-09-26; First posted 2020-10-06 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Major Depressive Disorder
Keywords: Psychotherapy; Mechanism of change; supportive-expressive treatment; Emotion-Focused Therapy; Psychodynamic psychotherapy; Insight; emotional processing
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double Blind (participants, outcome assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supportive-Expressive (Experimental): Participants will receive supportive-expressive treatment for 16 weeks.
  Interventions: Behavioral: Supportive-expressive treatment
- Emotion-Focused (Experimental): Participants will receive Emotion-Focused treatment for 16 weeks.
  Interventions: Behavioral: Emotions-Focused treatment

INTERVENTIONS:
Behavioral: Supportive-expressive treatment — Sixteen weeks of a time-limited psychodynamic therapy adapted for depression that includes the use of expressive techniques, such as interpretation, confrontation, clarification and the use of supportive techniques, such as affirmation and empathic validation. This treatment postulates insight as its core mechanism of change.
  Arms: Supportive-Expressive
Behavioral: Emotions-Focused treatment — Sixteen weeks of a brief experiential therapy for depression that combine client-centered relational elements (unconditional positive regard, congruence, and empathy) with marker-guided experiential interventions designed to facilitate and deepen emotional processing and emotion regulation.
  Arms: Emotion-Focused

SUMMARY:
This study will explore the mechanisms of change that are activated when individuals receive a treatment that targets their weakness and the mechanisms activated when the treatment capitalize on their strength. Patients will be assigned to one of two types of psychotherapies in treating people with a major depression disorder, expressive-supportive vs. emotion-focused treatment. Their ability to benefit from treatment based on their pre-treatment levels of insight and emotional processing will be examined. This is a four-month protocol, with a 2 year follow up period.

DETAILED DESCRIPTION:
One hundred and twenty-four patients suffering from major depressive disorder will be randomized to participate in 16 sessions of either supportive-expressive therapy or emotion-focused therapy. The two treatments are theorized to differ in their main mechanism of change: supportive-expressive therapy places emphasis on insight as its main mechanism of change, and emotion-focused therapy places emphasis on emotional processing as its main mechanism of change. Both can serve as strength- or weakness-focused treatments, based on the patient's baseline levels of insight and emotional processing. Importantly, this study will employ multiple complementary methods, which will include session-by-session self-report questionnaires from both patient and therapist, as well as interdisciplinary measures based on hormonal and acoustic measures, cognitive tasks, clinician interviews, and behavioral coding systems to complement the self-report measures. In addition, prior the beginning of treatment patients will complete diaries via mobile survey application. The findings will contribute to the research on personalized mechanisms of change and can help clinicians focus on more efficient treatment delivery, adapted to given subpopulations of patients, according to their strengths and weaknesses. If a mechanism most likely to stimulate change for a subpopulation is identified, a corresponding treatment can be chosen that is most likely to activate that particular mechanism and by that improve the rate of patients' respondent to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Meeting major depressive disorder diagnostic criteria using the structured clinical interviews for Diagnostic and Statistical Manual of Mental Disorders-5 and scoring more than 14 on the 17-item Hamilton rating scale for depression at two evaluations (one week apart) (Hamilton, 1967).
* If on medication, patients' dosage must be stable for at least three months prior to entering the study, and they must be willing to maintain stable dosage for the duration of treatment
* Age between 18 and 65
* Hebrew language fluency
* Provision of written informed consent.

Exclusion Criteria:

* Current risk of suicide or self-harm
* current substance abuse disorders
* current or past schizophrenia or psychosis, bipolar disorder, or severe eating disorder requiring medical monitoring
* history of organic mental disease
* currently in psychotherapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2020-11-29 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Weekly change in Hamilton rating scale for depression (HRSD) | up to 16 weeks.
  A 17-item clinically administered measure assessing the severity of depression. Higher scores indicate worse outcome.

SECONDARY OUTCOMES:
Weekly change in Beck Depression Inventory (BDI) | up to 16 weeks
  A 21-item, self-rated scale that evaluates key symptoms of depression. Higher scores indicate worse outcome.
Weekly change in Outcome Questionnaire (OQ) | up to 16 weeks
  A 30 items self-report measure designed to assess patient therapy outcomes on three primary dimensions: (a) subjective discomfort, (b) interpersonal relationships, and (c) social role performance. Higher scores indicate worse outcome.
Trajectories of change in Inventory of Interpersonal Problems (IIP-32) | At intake and 6 times during the treatment (weeks 1, 2, 4, 8, 12, 16)
  A 32-item self-report measure designed to assess interpersonal problems. Each item is rated in terms of how distressing the problem is for the individual on a scale ranging from 0 (not at all) to 4 (extremely). Higher scores indicate worse outcome.
trajectories of change in Quality of Life Enjoyment and Satisfaction- Short Version (Q-LES-Q) | At intake and 6 times during the treatment (weeks 1, 2, 4, 8, 12, 16)
  Quality of Life Enjoyment and Satisfaction Scale. Higher scores indicate better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Haifa, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No
Data will not be shared due to ethical reasons.

REFERENCES:
- [Derived] Zilcha-Mano S, Shahar B, Fisher H, Dolev-Amit T, Greenberg LS, Barber JP. Investigating patient-specific mechanisms of change in SET vs. EFT for depression: study protocol for a mechanistic randomized controlled trial. BMC Psychiatry. 2021 Jun 2;21(1):287. doi: 10.1186/s12888-021-03279-y. PMID 34078324